CLINICAL TRIAL: NCT04019509
Title: The Influence of Different Thyroid Autoantibodies on Thyroid Function and Pregnancy Outcome After Assisted Reproductive Technology
Acronym: TgAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Valerie Uvin, MD, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: TgABstudy Brussels
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Fertility Disorders; Thyroid Dysfunction
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tg AB positive, TPO AB negative (Active Comparator): Includes patients with only anti-thyroglobuline autoantibodies present and no anti-thyreoperoxydase antibodies at start of fertility treatment.
  Interventions: Diagnostic Test: blood test; Other: follow up treatment outcome
- Tg AB negative, TPO AB negative (Active Comparator): Includes patients without thyroid autoantibodies at start of fertility treatment
  Interventions: Diagnostic Test: blood test; Other: follow up treatment outcome
- Tg AB positive, TPO AB positive (Active Comparator): Includes patients with anti-thyroglobuline autoantibodies and anti-thyreoperoxydase antibodies at start of fertility treatment.
  Interventions: Diagnostic Test: blood test; Other: follow up treatment outcome

INTERVENTIONS:
Diagnostic Test: blood test — blood test for thyroid antibodies and thyroid function (TSH, FT4)
Other: follow up treatment outcome — questionnaire for treatment outcome: pregnancy, no pregnancy, miscarriage, delivery

SUMMARY:
The influence of thyroid autoantibodies on thyroid function in pregnancy after fertility treatment is not well known.

The objectives of the present study are:

1. To monitor the course of thyroid function during pregnancy and to compare between women with and without thyroid autoantibodies.
2. Compare pregnancy outcome between women with and without thyroid antibodies

DETAILED DESCRIPTION:
Thyroid autoantibodies and / or abnormal thyroid function are associated with fertility problems.

A possible explanation for this is, an influence of thyroid autoantibodies on the functioning of the thyroid gland. It is therefore recommended to check thyroid gland function and for the presence of autoantibodies before pregnancy. In general, 2 types of thyroid autoantibodies are known: anti-thyreoperoxidase autoantibodies and anti-thyroglobulin autoantibodies.

In case of abnormal thyroid function, treatment is sometimes necessary in regards to fertility. The risk of abnormal thyroid function is increased in women with thyroid autoantibodies during pregnancy. Therefore, thyroid function is regularly monitored during pregnancy in women with thyroid antibodies. The influence of thyroid autoantibodies on thyroid function in pregnancy after fertility treatment is not well known.

The objectives of the present study are:

1. To monitor the course of thyroid function during pregnancy and to compare between women with and without thyroid autoantibodies.
2. Compare pregnancy outcome between women with and without thyroid antibodies

ELIGIBILITY:
Inclusion Criteria:

* first cycle of assisted reproductive technology with follow up of thyroid function at the Universitair Ziekenhuis Brussel
* age >= 18 and <= 36 years
* body mass index between 18 and 35

Exclusion Criteria:

* Patients with clinical thyroid dysfunction
* Patients being treated with levothyroxine or antithyroid drugs
* Patients being treated with glucocorticosteroids
* Patients undergoing in vitro maturation or preimplantation genetic testing.
* Poor responders during IVF/ICSI stimulation, using the Bologna criteria

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
thyroid fonction | 12 months
  TSH, FT4 evolution during pregnancy
cumulative delivery rate | 12 months
  live birth delivery after IVF stimulation

SECONDARY OUTCOMES:
cumulative pregnancy rate | 12 months
  pregnancy rate after IVF stimulation
miscarriage rate | 12 months
  miscarriage rate after IVF stimulation

CONTACTS AND LOCATIONS:
Overall Officials: valerie uvin, md, Principal Investigator — UZ Brussels
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided